CLINICAL TRIAL: NCT06580873
Title: Evaluation of Switch to Dolutegravir/Lamivudine (DTG/3TC) From Current Suppressive Antiretroviral Therapy in People Living With HIV (PLWH) Receiving Opioid Agonist Therapy (OAT)
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Saskatchewan Health Authority - Regina Area (Other)
Collaborators: ViiV Healthcare (Industry)
Responsible Party: Principal Investigator, Alexander Wong, MD, Principal Investigator, Dr. Alexander Wong, Saskatchewan Health Authority - Regina Area
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REB-24-04
Record Dates: First submitted 2024-08-28; First posted 2024-08-30 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2024-08

CONDITIONS: HIV-1-infection; Opioid Use Disorder
Keywords: Antiretroviral Therapy
MeSH Terms: conditions — Opioid-Related Disorders | interventions — dolutegravir; Lamivudine

STUDY DESIGN:
Intervention Model Description: This study is a single-arm, open-label, prospective interventional cohort study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment Arm (Experimental): Switch to Dolutegravir/Lamivudine ("DOVATO") from current suppressive antiretroviral therapy in people living with HIV-1 receiving opioid agonist therapy.
  Interventions: Drug: DOVATO

INTERVENTIONS:
Drug: DOVATO — HIV-1 medication
  Other Names: Dolutegravir/Lamivudine

SUMMARY:
The goal of this clinical trial is to determine the efficacy of Dolutegravir/Lamivudine (DTG/3TC), or "Dovato", in virally-suppressed (HIV-1 RNA < 200 copies/mL) individuals receiving opioid agonist therapy such as methadone, buprenorphine, slow-release morphine, after switching from their current suppressive antiretroviral therapy (ART).

The main questions this trial seeks to answer are:

1. whether people living with HIV-1 (PLWH) on opioid agonist therapy (OAT) remain virally suppressed after switching to DTG/3TC from their current suppressive ART 48 weeks post-switch;
2. the number and type of adverse events (AEs) and serious adverse events (SAEs) attributable to DTG/3TC as documented per standard process at each study visit, and any discontinuations of DTG/3TC due to AEs and SAEs as determined by the study investigator;
3. the number of dosing changes in OAT attributable to DTG/3TC as determined by the study investigator and documented as per standard progress at each study visit;
4. the number of persons with any recreational or non-prescribed substances in their urine drug screens who remain virally suppressed (HIV-1 RNA < 200 copies/mL) at 48 weeks post-switch from current suppressive ART to DTG/3TC;
5. any change from baseline values (i.e., day 0) to 48 weeks post-switch from current suppressive ART to DTG/3TC of serum creatinine and non-fasting lipid parameters;
6. any change from baseline value (i.e., day 0) to 48 weeks post-switch from current suppressive ART to DTG/3TC in HIV Treatment Satisfaction Questionnaire (Status) (HIVTSQs) scores;
7. the number of persons who remain virally suppressed (HIV RNA < 200 copies/mL) at 48 weeks post-switch from current suppressive ART to DTG/3TC in conjunction with differing levels of adherence to DTG/3TC, and;
8. the number of persons who experience symptoms of opioid withdrawal or overdose per standardized survey or by self-report (e.g., overdose events)

During the course of the study, participants will complete:

* A set of questionnaires
* Blood draws
* A review of adverse events and concomitant medications
* ECG scans at screening and 48 weeks
* Urine drug screening
* Physical exams
* Review of alcohol consumption

DETAILED DESCRIPTION:
This study proposes to fill several important knowledge gaps regarding the safety and efficacy of switching to Dolutegravir/Lamivudine (DTG/3TC) in people living with HIV-1 (PLWH) on opioid agonist therapy (OAT) receiving care at the Infectious Diseases Clinic. As of this time, the Investigators are unaware of any real-world studies on the use of DTG/3TC in PLWH who are on OAT, PLWH using substances like fentanyl and crystal methamphetamine, or those of Indigenous ethnicity.

Additionally, clinical data on the use of DTG/3TC in young females is limited. The Infectious Diseases Clinic is well positioned to help further the understanding of real-world use of DTG/3TC among these understudied populations. With the inherent unpredictable adherence to current ART in PLWH receiving OAT, this study offers an opportunity to improve understanding of the real-world barrier to resistance of DTG/3TC in this clinical setting. The Principal Investigator proposes a single-arm, open-label, prospective interventional cohort study to evaluate the efficacy, and safety of switch to DTG/3TC from current suppressive ART in PLWH receiving OAT.

ELIGIBILITY:
Inclusion Criteria:

* Male and females, 18 years or older
* HIV-1 infected
* Prescribed a combination antiretroviral therapy (cART) regimen that may include any Department of Health and Human Services (DHHS) recommended or alternative regimens, which the treating physician considers is appropriate for their patient, except Dolutegravir/Lamivudine (DTG/3TC), or with DTG and 3TC as separate components of a single ART regimen at any point previously
* HIV-1 RNA < 200 c/mL at screening and at least 3 months prior to screening
* CD4 ≥ 200 cells/mL at screening
* Prescribed opioid agonist therapy (OAT) with oral methadone, sublingual buprenorphine, subcutaneous buprenorphine, slow-release oral morphine, or any combination thereof for at least 3 months prior to screening and deemed stable on OAT by the investigator
* Ability to remain adherent to medications and study protocol as per investigator opinion
* Must be willing and able to understand the requirements of study participation and provide signed and dated written informed consent prior to screening

Exclusion Criteria:

* Co-infection with hepatitis B (HBsAg positive). Individuals who are negative for HBsAg and anti-HBs but positive for hepatitis B core antibody (anti-HBc) will be excluded if they have detectable HBV DNA (i.e. greater than 10 IU/mL).
* History or presence of allergy to any component of DTG/3TC
* Documented or suspected resistance to any component of DTG/3TC
* Tuberculosis infection requiring treatment
* Concomitant use of drugs with contraindication or unmanageable drug interactions with any component of DTG/3TC
* Alanine transferase (ALT) greater than 5 times the upper limit of normal (ULN), or ALT greater than 3 times the ULN and bilirubin greater than 1.5 times the ULN (with >35% direct bilirubin)
* Has an estimated glomerular filtration rate (eGFR; by MDRD equation) < 30 mL/min/1.73m2
* Severe hepatic impairment (Class C or greater) by Child-Pugh classification
* Is pregnant, planning to get pregnant, or lactating
* Involved in any other interventional HIV study during the study period
* Has any reason, in the opinion of the investigator, which would make the candidate inappropriate for participation in an investigative study involving oral medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-09-30 (Estimated); Primary Completion 2026-05-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Number of people living with HIV-1 on opioid agonist therapy (OAT) that remain virally suppressed 48 weeks post-switch to Dolutegravir/Lamivudine (DTG/3TC) | Assessed at 48 weeks post-switch.
  The primary outcome assessed in the study is the number of individuals on OAT that remain virally suppressed (HIV RNA < 200 copies/mL) 48 weeks after switching from their current suppressive antiretroviral therapy (ART) to DTG/3TC.

SECONDARY OUTCOMES:
Changes in dosing of DTG/3TC | Through study completion, an average of 1 year.
  Number and type of adverse events (AEs) and serious adverse events (SAEs) attributable to DTG/3TC as documented per standard process at each study visit, and any discontinuations of DTG/3TC due to AEs and SAEs as determined by the study investigator.
Changes in dosing of OAT | Through study completion, an average of 1 year.
  Number of dosing changes in OAT attributable to DTG/3TC as determined by the study investigator and documented as per standard progress at each study visit.
Evidence of recreational drug use while maintaining suppression | Assessed at 48 weeks post-switch.
  The number of persons with any recreational or non-prescribed substances in their urine drug screens who remain virally suppressed (HIV-1 RNA < 200 copies/mL) at 48 weeks post-switch from current suppressive ART to DTG/3TC.
Changes in serum creatinine and non-fasting lipids | Assessed at 48 weeks post-switch.
  Change from baseline values (i.e., day 0) to 48 weeks post-switch from current suppressive ART to DTG/3TC of serum creatinine and non-fasting lipid parameters.
Change in HIV-1 Treatment Satisfaction Questionnaire (status) (HIVTSQs) scores | Assessed at 48 weeks post-switch.
  Change from baseline value (i.e., day 0) to 48 weeks post-switch from current suppressive ART to DTG/3TC in HIVTSQs scores, ranging from 0 to 60, with 0 being the least satisfied with current HIV-1 treatment, and 60 being the most satisfied.
Measurement of total adherence to DTG/3TC based on viral suppression | Assessed at 48 weeks post-switch.
  The number of persons who remain virally suppressed (HIV-1 RNA < 200 copies/mL) at 48 weeks post-switch from current suppressive ART to DTG/3TC in conjunction with differing levels of adherence to DTG/3TC.
Assessment of withdrawal symptoms or overdose | Through study completion, an average of 1 year.
  The number of persons who experience symptoms of opioid withdrawal or overdose per standardized survey or by self-report (e.g., overdose events).

CONTACTS AND LOCATIONS:
Locations (1):
- Saskatchewan Health Authority, Regina, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: No